CLINICAL TRIAL: NCT06702488
Title: The Efficacy of Dexmedetomidine and Magnesium Sulfate in Cognitive Dysfunction
Brief Title: Dexmedetomidine and Magnesium Sulfate in the Reduction Cognitive Dysfunction in Geriatrics
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Professor, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R577
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Mental Disorder
Keywords: Post-operative cognitive dysfunction
MeSH Terms: conditions — Mental Disorders | interventions — Dexmedetomidine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The dexmedetomidine (Active Comparator): 29 patients will receive a bolus dose of dexmedetomidine (0.5 μg kg-1) over 10 minutes before induction followed by an infusion (0.3 μg kg-1 h-1), which will be discontinued at the skin closure.
  Interventions: Drug: dexmedetomidine
- The magnesium sulfate (Active Comparator): 29 patients will receive 20 mg/kg as loading dose over 10 minutes before induction then maintenance dose 5 mg/kg/hour, which will also be discontinued at the skin closure
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — 20 mg/kg as a loading dose over 10 minutes before induction then a maintenance dose of 5 mg/kg/hour, which will also be discontinued at the skin closure.
  Other Names: magnesium sulfate

SUMMARY:
Magnesium sulfate is considered a neuroprotective drug and has been studied in various applications. Recently, it has drawn the attention of anesthesiologists, resulting in numerous publications about its role in anesthesiology.

Magnesium sulfate is suggested to exert its neuroprotective effect by preventing excitotoxicity. in the clinical setting, intraoperative magnesium sulfate attenuated POCD. Furthermore, postoperative emergence agitation was significantly reduced in pediatric patients who received intraoperative magnesium sulfate during adenotonsillectomy.

The aim of this study The aim of this work is to compare the protective effect of intraoperative dexmedetomidine with magnesium sulfate against developing POCD and to study their effect on serum level of CRP; the marker of neuronal degeneration.

DETAILED DESCRIPTION:
Post-operative cognitive dysfunction (POCD) in the elderly, defined as alteration either in thinking and/or impaired higher mental functions following surgery and anesthesia.

POCD should be seriously concerned in elderly people during induction of general anesthesia because of its high overall incidence rate (25.8% at one week, 9.9% after 3 months) with increasing the risk for it as the age advances due to physiologic changes that occurs, such as greater sensitivity to anesthetic drugs, higher drug concentrations at central nervous system receptors .

The etiology and pathogenesis of POCD following general anesthesia has gained much attention in the last years. recent research reveals a significant postoperative elevation of the marker of neuronal degeneration; S100β protein.S100β protein is an acidic calcium binding protein, found in astrocytes and schwann cells. Physiological serum levels of S100β protein are low, but in the early stages of neuronal injury, S100β is released into the blood. evidence suggested that overexpressed S100B can promote Aβ generation from amyloid precursor protein.The increased Aβ and amyloid precursor protein are known to be associated with cognitive impairment.consequently, postoperative elevation of S100β can be considered one of the possible mechanisms involved in the etiopathogenesis of POCD.

Dexmedetomidine have recently become prominent due to their increased use in anaesthetic and critical care practice for sedation and analgesia. dexmedetomidine suppress the inflammatory markers that are usually elevated in the post-surgical period, as well as neuronspecific markers of inflammation like neuron specific enolase (NSE) and S-100β, compared to controls Dexmedetomidine, a dextro-enantiomer of medetomidine and a highly selective a2 adrenoreceptor agonist, has sedative, analgesic, and sympatholytic properties, thereby reducing the requirement for anesthetic agents. a2 adrenergic receptors are abundant in the dorsal noradrenergic bundles, locus coeruleus, and frontal lobe, which are crucial for cognitive function and selective attention. Zhang et al. reported that a 0.5 μg kg-1 loading dose over 10 minutes followed by an infusion dose of 0.5 μg kg-1 h-1 in elderly patients undergoing laparoscopic surgery under general anesthesia for colorectal cancer provided neuroprotection regarding the reduced incidence of POCD and neuroinflammatory marker levels. A meta-analysis also found that dexmedetomidine during surgery suppressed inflammatory cytokines, particularly IL-1 and IL-6, perioperatively and helped preserve cognitive functions in the elderly . It has been reported that postoperative elevation of peripheral C-reactive protein (CRP) and interleukin 6 concentrations is associated with higher risks of postoperative delirium.Interestingly, the authors also found that increased preoperative concentrations of CRP and interleukin 6 are also associated with an increased risk of postoperative delirium, thus supporting the hypothesis that preoperative pathologies may also contribute to the risk of subsequent postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I, II and ⅠⅠⅠ
* patients undergoing open abdominal surgery under general anesthesia

Exclusion Criteria:

* Elderly patients with preoperative MoCA Score below 26.
* Operation time more than 4 hours to prevent excessive dosage of magnesium sulfate.
* BMI > 35 kg m-2

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
the incidence of Post Operative Cognitive Dysfunction | 24 hours postoperative
  Post Operative Cognitive Dysfunction

SECONDARY OUTCOMES:
CRP levels and their correlation with POCD | 24 hours of postoperative
  CRP levels and their correlation with POCD

CONTACTS AND LOCATIONS:
Locations (1):
- Dexmedetomidine, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No
no plan to share

REFERENCES:
- [Result] BEDFORD PD. Adverse cerebral effects of anaesthesia on old people. Lancet. 1955 Aug 6;269(6884):259-63. doi: 10.1016/s0140-6736(55)92689-1. No abstract available. PMID 13243706